CLINICAL TRIAL: NCT00989547
Title: Transfusion of Autologous Umbilical Cord Blood to Reverse Hyperglycemia in Children With Type 1 Diabetes - A Pilot Study.
Brief Title: Cord Blood Infusion for Type 1 Diabetes Mellitus (T1DM)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 593
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Type 1 Diabetes; Children
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Other: Umbilical Cord Blood VITA 34
- B (No Intervention)

INTERVENTIONS:
Other: Umbilical Cord Blood VITA 34 — Intervention type: Autologous Umbilical Cord Blood Transfusion
  Arms: A

SUMMARY:
Type 1 diabetes (T1D) is still associated with tremendous morbidity and premature mortality.

Patients require multiple daily insulin injections throughout their lives as well as close monitoring of their diet and blood sugar levels to prevent complications. Unfortunately, there is presently no permanent cure for diabetes. Whole pancreas or islet cell transplantation is available only to a very limited number of patients and necessitates potential lifelong immunosuppressive therapy. Autologous stem cell transplants have been used successfully for ALL (acute lymphoblastic leukemia), AML (acute myeloblastic leukemia) and for the treatment of a variety of cancers including breast cancer and neuroblastomas, and more recently for the treatment of autoimmune disorders such as multiple sclerosis (MS), lupus-like disease, and rheumatic disorders. Recently it was shown that bone marrow-derived stems cells transplanted into diabetic mice led to reduced hyperglycemia within 7 days after transplantation and was sustained until they were sacrificed at 35 days post-transplantation. The investigators' goal is to transfuse autologous umbilical cord blood into 23 children (Germany 10 and 20 Controls) with T1D in an attempt to regenerate pancreatic islet insulin producing beta cells and improve blood glucose control. As secondary goals, the investigators aim to track the migration of transfused cord blood stem and study the potential changes in metabolism/immune function leading to islet regeneration.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of T1D and have stored umbilical cord blood (10 patients sought) at the cord bank Vita 34.
* TID diagnosis will be defined as having a clear history of polydipsia, polyphagia, polyuria, and weight loss consistent with a clinical diagnosis, diagnosis will mot be based solely upon the presence of autoantibodies.
* Cord blood meets all selection and testing criteria (see below).
* Normal screening values for CBC, Renal function and electrolytes (BMP).
* Willing to comply with intensive diabetes management
* Not younger than 1 year of age

Exclusion Criteria:

* Have complicating medical issues that would interfere with blood drawing or monitoring.
* Require chronic use of steroids or other immunosuppressive agents for other conditions.
* Cord Blood with viability < 50%.
* Positive infectious disease markers from mothers blood or cord at time of collection (See below for details).
* Any evidence of illness on planned infusion date (i.e. fever >38.5 C, vomiting, diarrhea, wheezing, or crackles).

Min Age: 1 Year | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-09; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
insulin production
  change in median area under the curve (AUC) for C-peptide (measure of insulin production) from baseline to 2 years during a 2h Mixed Meal Tolerance Test was used as the primary outcome measure and was reported in ng/mL/120 minutes.

SECONDARY OUTCOMES:
Insulin Dose, Autoantibody levels, T-cell functional response assays, Cytokine levels
  Insulin Dose, Autoantibody levels, T-cell functional response assays, Cytokine levels

OTHER OUTCOMES:
glycated hemoglobin (HbA1c)

CONTACTS AND LOCATIONS:
Locations (1):
- Forschergruppe Diabetes der Technischen Universität, München, Bavaria, Germany